CLINICAL TRIAL: NCT01429129
Title: Randomized Controlled Trial of Mailed Nicotine Replacement Therapy to Canadian Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 029/2011
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Smoking
Keywords: Smoking; Nicotine; Nicotine Replacement Therapy; Nicotine Patch; Nicoderm; Mass Distribution; Tobacco Control; Randomized Controlled Trial
MeSH Terms: conditions — Smoking | interventions — Nicotine Replacement Therapy; Nicotine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Replacement Therapy (Experimental)
  Interventions: Drug: Nicotine replacement therapy
- Control (No Intervention)

INTERVENTIONS:
Drug: Nicotine replacement therapy — Nicotine transdermal patches as per product monograph
  Other Names: Nicoderm
  Arms: Nicotine Replacement Therapy

SUMMARY:
This study will examine the efficacy of mailed distribution of free Nicotine Replacement Therapy to smokers. Telephone numbers will be randomly selected from across Canada in order to recruit adult smokers interested in completing a smoking survey and willing to be interviewed again in 8 weeks and 6 months time. Study participants will be asked about their smoking history and a hypothetical question: would they be interested in receiving the nicotine patch if this were to be provided to them free of charge? Participants expressing interest will be randomly assigned to one of two groups. One group will be offered the opportunity to actually receive a program of 5 weeks of the nicotine patch for free right away and the other group will not be offered the free nicotine patches. The proportions of smokers in the two groups who quit smoking by the 6-month interview will be compared.

DETAILED DESCRIPTION:
Tobacco smoking is the leading cause of preventable death. Considerable public health efforts are ongoing Canada-wide to reduce the prevalence of smoking in the general population. From 1985 to 2005, smoking rates among adults reduced from 35% to 19%. However, since that time, this steady rate of decline plateaued at around 18-19%. What else can be done to continue to significantly reduce the number of smokers at the population level? One option is to translate interventions that have demonstrated clinical efficacy into population level initiatives. Nicotine Replacement Therapy (NRT) has a considerable research base demonstrating its efficacy. Public health initiatives are underway to distribute NRT widely through mass distribution efforts. For example, over 58,000 NRT treatments have been distributed in the province of Ontario alone, and other provinces in Canada are considering adopting mass distribution procedures. However, one important question remains unanswered - do smoking cessation programs that involve mass distribution of free NRT work? Preliminary evidence consisting of before-after smoking status data from participants of mass NRT campaigns yielded promising results. However, such data cannot be used to make causal statements about the impact of NRT distribution. To answer this question, a randomized controlled trial is required.

A single blinded, panel survey design with random assignment to an experimental and a control condition will be used in this study. A two-stage recruitment process will be employed, in the context of a general population survey with two follow-ups (8 weeks and 6 months). Random digit dialing of Canadian home telephone numbers will identify households with adult smokers who are willing to take part in a smoking study that involves three interviews, with saliva collection for 3-HC/cotinine ratio measurement at baseline and saliva cotinine verification at 8-week and 6-month follow-ups.

As part of the baseline survey, eligible subjects will be identified for the second recruitment - randomization of smokers into experimental and control conditions to receive versus not receive nicotine patches. Eligibility will be determined by a series of questions regarding hypothetical interest in nicotine patches to quit smoking (including willingness to have nicotine patches sent to their home) and having no contraindications for using NRT. A randomized half of the eligible subjects will be assigned to the experimental condition and asked for their permission to have nicotine patches sent to their home. Subjects will be followed-up at 8 weeks and 6 months. Subjects in the control condition will not be offered nicotine patches. Interviewers will be blind to subjects' condition because they will be using computer assisted telephone interviewing (CATI) technology and as the first parts of the 8-week and 6-month follow-ups are identical for experimental and control conditions, they will not know the intervention condition to which a subject belongs until questions specific to the use of NRT are asked near the end of the surveys (i.e., after the primary outcome measures are assessed).

The primary hypothesis is that subjects who receive nicotine patches at baseline will display significantly higher quit rates (as assessed by 30 day point prevalence of abstinence from tobacco) at 6-month follow-up as compared to subjects who do not receive nicotine patches at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Current daily smokers who smoke 10 or more cigarettes per day
* Interested in being involved in a smoking study
* Willing to be interviewed at baseline, 8 weeks and 6 months after
* Willing to provide a saliva sample for cotinine analysis at each time point
* Interest in using nicotine patch to quit smoking
* Intent to use nicotine patch within one week of receiving it
* Willing to have nicotine patch sent to their home

Exclusion Criteria:

* Have a medical condition that would would make participation medically hazardous as determined by the list of contraindications for NRT outlined in the CPS and the NRT package insert
* Pregnant, intending on becoming pregnant, or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 6 month follow-up

SECONDARY OUTCOMES:
Smoking cessation | 8 week follow-up
Reduction in smoking since baseline | past 6 months
Compliance with course of nicotine patches provided | past 6 months
Purchase and use of NRT and smoking cessation aids | past 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kushnir V, Selby P, Zawertailo L, Tyndale RF, Leatherdale ST, Cunningham JA. Long-term effectiveness of mailed nicotine replacement therapy: study protocol of a randomized controlled trial 5-year follow-up. BMC Public Health. 2017 Jul 18;18(1):28. doi: 10.1186/s12889-017-4586-z. PMID 28720080
- [Derived] Kushnir V, Sproule BA, Cunningham JA. Impact of large-scale distribution and subsequent use of free nicotine patches on primary care physician interaction. BMC Public Health. 2017 Jul 11;18(1):4. doi: 10.1186/s12889-017-4548-5. PMID 28693456
- [Derived] Kushnir V, Sproule BA, Zawertailo L, Selby P, Tyndale RF, Leatherdale ST, Cunningham JA. Impact of self-reported lifetime depression or anxiety on effectiveness of mass distribution of nicotine patches. Tob Control. 2016 Sep;26(5):526-533. doi: 10.1136/tobaccocontrol-2016-052994. Epub 2016 Aug 19. PMID 27543563
- [Derived] Cunningham JA, Kushnir V, Selby P, Tyndale RF, Zawertailo L, Leatherdale ST. Effect of Mailing Nicotine Patches on Tobacco Cessation Among Adult Smokers: A Randomized Clinical Trial. JAMA Intern Med. 2016 Feb;176(2):184-90. doi: 10.1001/jamainternmed.2015.7792. PMID 26809849
- [Derived] Cunningham JA, Leatherdale ST, Selby PL, Tyndale RF, Zawertailo L, Kushnir V. Randomized controlled trial of mailed Nicotine Replacement Therapy to Canadian smokers: study protocol. BMC Public Health. 2011 Sep 28;11:741. doi: 10.1186/1471-2458-11-741. PMID 21955930